CLINICAL TRIAL: NCT03031210
Title: Treatment of Non-severe Community Acquired Pneumonia With Twice Daily Compared to Thrice Daily Regimen- A Non-inferiority Pragmatic Randomized-controlled Trial.
Brief Title: Twice Daily Treatment With Amoxicillin for Non-severe Community Acquired Pneumonia.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, Principal investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BID pneumonia
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Community-acquired Pneumonia
Keywords: Non-severe community-acquired pneumonia; Amoxicillin treatment; Twice daily antibiotic regimen
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Twice a day regimen (Experimental): Patients will received a prescription of amoxicillin (90mg/kg/day) divided in two doses daily.
  Interventions: Drug: Amoxicillin
- Thrice a day regimen (Active Comparator): Patients will received a prescription of amoxicillin (90mg/kg/day) divided in three doses daily.
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — (90 mg/kg/day) twice daily
  Other Names: Amoxil

SUMMARY:
The aim of this study will be to evaluate whether a twice-daily antibiotic regimen is non-inferior to a thrice-daily regimen for the treatment of non-severe community acquired pneumonia in children presenting at a paediatric Emergency Department (ED).

DETAILED DESCRIPTION:
A single-center, non-blinded, pragmatic, randomized-controlled, non-inferiority clinical trial will be conducted in an urban, university-affiliated, tertiary care pediatric hospital ED. All patients three months old to 18 years of age who had symptoms and signs suggestive of non-severe community acquired pneumonia based on respiratory complaints and a pulmonary infiltrate identified by trained paediatricians or emergency physicians will be eligible to the present study. Study participants will be randomly allocated to receive either amoxicillin (90mg/kg per day) in twice or thrice daily regimen. Primary outcome will be treatment failure within 10 days of enrolment as defined by hospitalisation, need for a change in antibiotic (persistence of fever at 72 hours, clinical deterioration, comorbid condition or development of serious adverse reactions) and death. ED revisits within 72 hours, second course of antibiotic and clinical recurrence rates will be evaluated in the follow-up assessments as well as percent of adverse events encountered, number of days missed (work, school or daycare), coverage vaccination rate, protocol adherence and patient and parental satisfaction. The primary analysis will use an intention-to-treat approach. Per-protocol analysis will also be carried to compare the failure rate. Accounting to a maximal 10% drop-off rate, a sample size of 685 participants per arm was calculated to have a power of 90% to identify a difference of ≤ 5% with an alpha value of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All patients 3 months to 18 years of age attending the pediatric ED and diagnosed with a non-severe pneumonia, will be considered for enrolment. More precisely, the following inclusion criteria will be required:

  1. Presence of respiratory symptoms (cough and/or dyspnea)
  2. Presence of signs of pneumonia (tachypnea, abnormal breath sounds, crackles)
  3. Presence of fever
  4. Positive chest radiography as interpreted by the treating physician

Exclusion Criteria:

* Any danger signs associated with pneumonia (severe indrawing, shock or severe dehydration, empyema, important pleural effusion, pulmonary abcess or pneumatocoele)
* History of anaphylactic or allergic reaction to penicillin or amoxicillin according to the treating physician.
* History of a serious nonimmunoglobulin E-mediated reactions (eg, Stevens-Johnson syndrome or toxic epidermal necrolysis) attributed to amoxicilin.
* Caregiver unable to provide consent (language barrier or lack of caregiver presence)
* Underlying unstable chronic illness (ie. cystic fibrosis, immune suppression, active tuberculosis, bronchiectasis or active pulmonary malignancies)
* Persistent/chronic pneumonia syndromes (with symptoms for >2 weeks), suspected by the physician to be caused by atypical pathogens, hospital- acquired pneumonia (been hospitalized within 2 weeks prior to enrolment), aspiration pneumonia or recurrent pneumonias.
* Any history of receiving amoxicillin within the past month
* Need hospitalisation for any other reasons (ie. persistent vomiting, severe life-threatening infection such as septicaemia or meningitis requiring intravenous antimicrobial agents)
* Previous participation in study

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1370 (Estimated)
Dates: Start 2017-06-11 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical failure within 10 days of enrolment | Day 10 (after enrolment)
  As a primary outcome, clinical failure will be defined by any of the following occurring within 10 days of enrolment:
  * Death or hospitalisation
  * A need for a change in antibiotic according to the treating physician. In our settings, common reasons to change antibiotic are:
    * Persistence of fever at 72h
    * Clinical deterioration:
      • Clinical deterioration will include the development of lower chest-wall indrawing, central cyanosis, stridor while calm, or danger signs as defined by: inability to drink or breastfeed, convulsions, persistent vomiting, lethargy, or unconsciousness at any time during a child's treatment.
    * Development of a comorbid condition such as a meningitis, bacteriemia, osteomyelitis or septic arthritis
    * Allergic reaction

SECONDARY OUTCOMES:
Emergency department revisit within 72 hours | 72 hours
  Return to the emergency department in the following 72 hours
Second course of antibiotic | 1 month
  Necessity of second course of antibiotics
Clinical recurrence | 1 month
  Another diagnosis of pneumonia
Adverse events | 10 days
  Any adverse event
Number of working days missed by caregivers or school/daycare days missed by patients | 1 month
  Total number of days missed by caregivers or school/daycare days missed by the parents
Patient's and parents satisfaction with the discharge instructions' provided and the ease of administration | 10 days
  Measured on a likert scale through a telephone survey

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Gravel, MD, Principal Investigator — Sainte-Justine Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No